CLINICAL TRIAL: NCT05923398
Title: Digital Interventions to Understand and Mitigate Stress Response: Process & Content Evaluation to Move From Feasibility (SRL-4) to Simulated Demonstration (SRL-6)
Brief Title: Digital Interventions to Understand and Mitigate Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Toronto Metropolitan University (Other); University of Toronto (Other); University of Ontario Institute of Technology (Other); Boston University (Other); University of Ottawa (Other); Western University, Canada (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-279
Record Dates: First submitted 2022-12-20; First posted 2023-06-28 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Distress, Emotional; Stress Response Among Nursing Professionals During the COVID-19; Stress Reaction; Acute
Keywords: Moral distress; Stress; Virtual Reality; Wearables; Web-based intervention; Nursing professionals; Nursing staff; Distress; COVID-19
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; COVID-19

STUDY DESIGN:
Intervention Model Description: Over approximately 3.5 months, each nursing professional will participate in the following:
  A) Undergo a virtual reality scenario to understand and reduce stress and moral distress related to difficult decision-making in complex moral situations during the COVID-19 pandemic.
  B) Use a web-based platform to measure stress, moral distress, and other mental health symptoms, as well as a commercial wearable device to collect physiological, sleep, and activity data to understand and examine the contribution of active and passive data to stress and moral distress.
  During analysis, once all passive and active data is collected we will create a personal digital phenotype profile (pDPP) based on the physiological data collected during a morally challenging situation in a virtual environment as well as the wearable and web-based data to help understand stress and moral distress at the individual level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): During the duration of the study, all participants will use the Digital Intervention Suite (a web-based component, a VR platform, and wearable device) to measure passive and active data, such as: psychological variables (e.g., moral distress, anxiety, and depression) and physiological variables (e.g., heart rate and sleep).
  Interventions: Behavioral: Digital Intervention Group

INTERVENTIONS:
Behavioral: Digital Intervention Group — Participants will use a Digital Intervention Suite composed of a virtual reality (VR) scenario, a web-based platform, and a wearable device to assess their stress response in near-real time and in a hypothetical stressful scenario.
  During the VR scenario, physiological signals such as Galvanic Skin Response (GSR), Electrocardiogram (ECG), Respiratory Independence (RI), and Photoplethysmography will be measured. Additionally, an educational intervention video on how to deal with stress and distress will be shown to participants. We will then request participants to practice the skills taught during the intervention video in the VR scenario.
  The wearable device (Oura Ring) will measure sleep, activity, readiness information, heart rate, heart rate variability, body temperature (delta), and respiratory rate. Additionally, the web-based platform will, through questionnaires, assess stress-related symptoms such as loneliness, anxiety, depression, and moral injury.

SUMMARY:
Stress, anxiety, distress, and burnout are exceptionally high among healthcare workers at the frontline of the COVID-19 pandemic. The understanding of factors underlying distress and resilience in complex workplace contexts is limited, and there are limited evidence-based interventions for stress and moral distress among frontline healthcare workers. The purpose of this study is to use a Digital Intervention Suite (a combination of Virtual Reality [VR], a web-based platform, and a wearable [Oura Ring]) to understand and reduce the experience of stress/distress faced by nursing professionals.

DETAILED DESCRIPTION:
The purpose of this study is to use a Digital Intervention Suite (a combination of Virtual Reality [VR], a web-based platform, and a wearable [Oura Ring]) to understand and reduce the experience of stress/distress faced by nursing professionals. This study involves participation in an in-person VR setup and the use of an app and a wearable device over the duration of the study (14+ weeks). The immersive VR component of the study involves a virtual experience of navigating a challenging workplace scenario to understand stress response and provide an overview of interventions that can be used to reduce workplace stress. Upon completion of the in-person VR visit, participants will continue to use the app and the wearable for the study duration to understand stress responses in their actual workplaces. Participants will have real-time access to their essential data on wellness collected through the app and wearable (e.g., sleep, activity, physiological signals, anxiety symptoms). The Digital Intervention Suite (combined use of these three components: VR, app, and wearable) is essential for a thorough understanding of stress and moral distress. This is a de-identified study, and the team will only have access to de-identified data for analysis at the end of the study.

ELIGIBILITY:
Inclusion criteria:

1. Registered nurses (RNs) or registered practical nurses (RPNs) who are currently employed at a healthcare institution in Ontario.
2. Ownership of a smartphone.

Exclusion criteria:

1. History of seizures (except febrile seizure).
2. Use of electronic medical devices (e.g., cardiac pacemakers, hearing aids, and defibrillators).
3. A score of ≥ 15 on the Generalized Anxiety Disorder (GAD-7) scale
4. A score of ≥ 20 on the Patient Health Questionnaire (PHQ-9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | Approximately 3.5 months
  The primary outcome will be the change in SUDS scores from (1) beginning to end of VR and (2) baseline to end of follow-up.
  The SUDS is an instrument (visualized as a fear thermometer) that ranges from scores of 0 to 100. It measures the intensity of emotions and other internal experiences, such as anxiety, anger, agitation, tension, and other painful emotions.
  Participants will complete SUDS before the VR scenario starts and once the VR scenario is over. Additionally, participants will complete the SUDS for a total of 8 times when in the VR scenario. Participants will also answer the SUDS using the web-based platform every week on Mondays, Thursdays, and Saturdays for approximately 3.5 months.
Moral Injury Outcome Scale (MIOS-4; 4 item scale) | Approximately 3.5 months
  The primary outcome will be the change in MIOS-4 scores from (1) beginning to end of VR and (2) baseline to end of follow-up.
  MIOS-4 is a short version of the MIOS-14. The 4 items have scores that range 0 (strongly disagree) to 4 (strongly agree); Total score ranges from 0 - 16.
  The MIOS is intended to measure the severity of moral injury outcomes as a result of a potentially morally damaging experience.
  Participants will complete the MIOS-4 during the VR scenario for a total of 8 times. Additionally, participants will answer the MIOS-4 using the web-based platform every week on Mondays and Thursdays for approximately 3.5 months.

SECONDARY OUTCOMES:
UCLA Loneliness Scale (3 item scale) | Approximately 3.5 months
  This secondary outcome will be the change in UCLA scores from baseline to end of follow-up.
  Short, 3-item scale. Item's scores range from 1 (hardly ever) to 3 (often) and total score ranges from 3 to 9. Higher scores indicate more severe loneliness symptoms.
  Participants will answer the UCLA-3 using the web-based platform every week on Mondays and Thursdays for approximately 3.5 months.
Generalized Anxiety Disorder Scale (GAD-7; 7 item scale) | Approximately 3.5 months
  This secondary outcome will be the change in GAD-7 scores from baseline to end of follow-up.
  The GAD-7 is a 7-item scale with each item's score ranging from 0 (not at all) to 3 (nearly everyday). Total score ranges from 0 to 21. Higher scores indicate more severe anxiety symptoms.
  Participants will answer the GAD-7 using the web-based platform every week on Saturdays for approximately 3.5 months.
Generalized Anxiety Disorder Scale (GAD-2; 2 item scale) | Approximately 3.5 months
  This secondary outcome will be the change in GAD-2 scores from baseline to end of follow-up.
  The GAD-2 only includes items 1 and 2 of the GAD-7. Each item's score ranges from 0 (not at all) to 3 (nearly everyday). Total score ranges from 0 to 6.
  Participants will answer the GAD-2 using the web-based platform every week on Mondays and Thursdays for approximately 3.5 months.
Patient Health Questionnaire (PHQ-9; 9 item scale) | Approximately 3.5 months
  This secondary outcome will be the change in PHQ-9 scores from baseline to end of follow-up.
  The PHQ-9 is a 9-item scale with each item's score ranging from 0 (not at all) to 3 (nearly every day). Total score ranges from 0 to 27. Higher scores indicate more severe depression symptoms.
  Participants will answer the PHQ-9 on Saturdays for approximately 3.5 months.
Patient Health Questionnaire (PHQ-2; 2 item scale) | Approximately 3.5 months
  This secondary outcome will be the change in PHQ-2 scores from baseline to end of follow-up.
  The PHQ-2 only includes items 1 and 2 of the GAD-9. Each item's score ranging from 0 (not at all) to 3 (nearly every day). Total score ranges from 0 to 6.
  Participants will answer the PHQ-2 using the web-based platform every week on Mondays and Thursdays for approximately 3.5 months.
Moral Injury Outcome Scale (MIOS-14; 22 item scale) | Approximately 3.5 months
  The primary outcome will be the change in MIOS-14 scores from (1) beginning to end of VR and (2) baseline to end of follow-up.
  MIOS-14 is a 22 item scale. Scores on the first 14 items range from 0 (strongly disagree) to 4 (strongly agree); total score ranges from 0 to 56. The other 8 items have scores that range from 0 (not at all) to 6 (extremely); total score ranges from 0 to 48.
  Participants will complete the MIOS-14 before the VR scenario starts and once the VR scenario is over. Additionally, participants will complete the MIOS-14 every Saturday for approximately 3.5 months.

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Bhat, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin J, Rueda A, Lee GH, Tassone VK, Park H, Ivanov M, Darnell BC, Beavers L, Campbell DM, Nguyen B, Torres A, Jung H, Lou W, Nazarov A, Ashbaugh A, Kapralos B, Litz B, Jetly R, Dubrowski A, Strudwick G, Krishnan S, Bhat V. Digital Interventions to Understand and Mitigate Stress Response: Protocol for Process and Content Evaluation of a Cohort Study. JMIR Res Protoc. 2024 May 6;13:e54180. doi: 10.2196/54180. PMID 38709554